CLINICAL TRIAL: NCT00047008
Title: A Phase III Trial of Concurrent Radiation and Chemotherapy for Advanced Head and Neck Carcinomas
Brief Title: Chemotherapy and Radiation Therapy With or Without Surgery in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0129; CDR0000257233; RTOG-H-0129
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard fractionation RT + cisplatin (Other): Standard fractionation radiation therapy with concurrent cisplatin followed by conventional surgery for select patients.
  Interventions: Drug: cisplatin; Radiation: Standard fractionation RT; Procedure: Conventional surgery for select patients
- Accelerated fractionation RT + cisplatin (Experimental): Accelerated fractionation radiation therapy by concomitant boost with concurrent cisplatin followed by conventional surgery for select patients.
  Interventions: Drug: cisplatin; Radiation: Accelerated fractionation radiation therapy; Procedure: Conventional surgery for select patients

INTERVENTIONS:
Drug: cisplatin — 100 mg/m^2 intravenously on days 1, 22
Radiation: Standard fractionation RT — Radiation will be delivered in 2 Gy per fraction, five fractions a week. The primary tumor and clinically/radiologically involved nodes will receive 70 Gy in 7 weeks and uninvolved nodes will receive 50 Gy in 5 weeks. The anterior lower neck field will be treated with 2 Gy per fraction at 3-cm depth to a total dose of 50 Gy.
  Arms: Standard fractionation RT + cisplatin
Radiation: Accelerated fractionation radiation therapy — Radiation to the initial target volume encompassing the gross and subclinical disease sites will be delivered in 1.8 Gy per fraction, five fractions a week to 54 Gy in 30 fractions over 6 weeks. At 32.4 Gy/18 Fx (i.e., latter part of week 4), the boost volume covering gross tumor and clinically/radiologically involved nodes will receive boost irradiation of 1.5 Gy/Fx as second daily fraction (at least 6 h interval) for a total of 12 treatment days (18 Gy total). The primary tumor and clinically/radiologically involved nodes will receive 72 Gy in 42 fractions over 6 weeks and uninvolved nodes will receive 54 Gy in 6 weeks. Clinically/radiologically negative posterior neck should receive a minimum dose of 50.4 Gy at 3 cm. The anterior lower neck field will be treated with 1.8 Gy per fraction at 3-cm depth to a total dose of 50.4 Gy in 28 fractions in 5.6 weeks.
  Arms: Accelerated fractionation RT + cisplatin
Procedure: Conventional surgery for select patients — Surgical removal (salvage resection) of the primary tumor should be performed if biopsy-proven cancer remains more than three months after completion of therapy. The nature of the surgical resection should be dictated by the extent of tumor at the initial evaluation. The operation should be conducted using accepted criteria for primary surgical treatment of the cancer.
  A planned neck dissection for patients with multiple neck nodes or with lymph nodes exceeding 3 cm in diameter (N2a, N2b, N3) is mandatory, regardless of the clinical and/or radiographic response. A neck dissection is required for patients with N1 disease if a palpable or worrisome radiographic abnormality persists in the neck six weeks after completion of therapy. Surgery should be performed within 2 weeks once the decision for neck dissection is made.

SUMMARY:
RATIONALE: Radiation therapy (RT) uses high-energy x-rays to damage tumor cells. Giving radiation therapy in different ways and combining it with chemotherapy before surgery may kill more tumor cells. It is not yet known which radiation therapy regimen combined with chemotherapy with or without surgery is more effective for head and neck cancer.

PURPOSE: Randomized phase III trial to compare two different radiation therapy regimens combined with cisplatin with or without surgery in treating patients who have stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with stage III or IV squamous cell carcinoma of the head and neck treated with conventional vs accelerated radiotherapy and concurrent cisplatin with or without surgical resection.

Secondary

* Compare local-regional control of disease and disease-free rates in patients treated with these regimens.
* Compare the acute and late toxicity of these regimens in these patients.
* Compare quality of life, perception of side effects, and performance status of patients treated with these regimens.
* Determine whether epidermal growth factor receptor and cyclo-oxygenase-2 expressions are independent prognostic markers in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor site (larynx vs other), nodal stage (N0 vs N1 or N2a or N2b vs N2c or N3), and Zubrod performance status (0 vs 1). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard fractionation radiotherapy 5 days a week for 7 weeks. Patients also receive cisplatin IV on days 1, 22, and 43.
* Arm II: Patients undergo accelerated fractionation radiotherapy 5 days a week for 3.5 weeks and then twice a day, 5 days a week, for 2.5 weeks. Patients also receive cisplatin IV on days 1 and 22.

Patients with biopsy-proven relapsed disease more than 3 months after completion of therapy undergo surgical resection of the primary tumor.

Quality of life is assessed at baseline, during one of the last 2 weeks of treatment, at 3 and 12 months, and then annually for 4 years.

Patients are followed at 6-8 weeks, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 720 patients (360 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx

  * Stage III or IV (T2, N2-3, M0 or T3-4, any N, M0)
* No metastases below the clavicle or more distant by clinical exam or radiology

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) no greater than 2 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 50 mL/min
* Calcium normal

Cardiovascular

* No symptomatic coronary artery disease (angina)
* No myocardial infarction within the past 6 months

Other

* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer
* No simultaneous primary tumors
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the head and neck except radioactive iodine therapy

Surgery

* No prior surgery to the primary tumor or nodes except diagnostic biopsy or nodal sampling of neck disease

  * No radical or modified neck dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2002-07 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phuc Felix Nguyen-Tan, MD, Principal Investigator — CHUM Hospital Notre Dame
Locations (195):
- United States (195):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Osborn, Scottsdale, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Saint Rose Hospital, Hayward, California
  - Cancer Care Consultants Medical Associates at Daniel Freeman Memorial Hospital, Inglewood, California
  - Valley Memorial Hospital, Livermore, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Highland General Hospital, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Radiological Associates of Sacramento Medical Group, Inc., Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Naval Medical Center - San Diego, San Diego, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida - Jacksonville, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Florida Shands Cancer Center, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Alexian Brothers Cancer Care Center, Elk Grove Village, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - St. John's Cancer Center at St. John's Medical Center, Anderson, Indiana
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center - Plymouth Campus, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Cancer Treatment Center at the Medical Center - Bowling Green, Bowling Green, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Cancer Center at Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - New Orleans Cancer Institute at Memorial Medical Center, New Orleans, Louisiana
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - South Suburban Oncology Center, Quincy, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Cancer Institute of Cape Girardeau, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Healthcare Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - John Smith, Jr./Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - LaFortune Cancer Center at St. John Health System, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cancer Center at Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Rappahannock General Hospital, Kilmarnock, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Community Memorial Health Center, South Hill, Virginia
  - North Star Lodge Cancer Center, Yakima, Washington
  - Washington Hematology - Oncology Specialists, Yakima, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Mary's Cancer Center at Columbia St. Mary's Hospital - Milwaukee Campus, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillison ML, Zhang Q, Jordan R, Xiao W, Westra WH, Trotti A, Spencer S, Harris J, Chung CH, Ang KK. Tobacco smoking and increased risk of death and progression for patients with p16-positive and p16-negative oropharyngeal cancer. J Clin Oncol. 2012 Jun 10;30(17):2102-11. doi: 10.1200/JCO.2011.38.4099. Epub 2012 May 7. PMID 22565003
- [Result] Wuthrick EJ, Zhang Q, Machtay M, et al.: The influence of institutional head and neck cancer (HNC) clinical trial accrual on overall survival (OS): An analysis of RTOG 0129. [Abstract] J Clin Oncol 30 (Suppl 15): A-5530, 2012.
- [Result] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Result] Ang K, Zhang Q, Wheeler RH, et al.: A phase III trial (RTOG 0129) of two radiation-cisplatin regimens for head and neck carcinomas (HNC): impact of radiation and cisplatin intensity on outcome. [Abstract] J Clin Oncol 28 (Suppl 15): A-5507, 2010.
- [Result] Gillison ML, Harris J, Westra W, et al.: Survival outcomes by tumor human papillomavirus (HPV) status in stage III-IV oropharyngeal cancer (OPC) in RTOG 0129. [Abstract] J Clin Oncol 27 (Suppl 15): A-6003, 2009.
- [Result] Ang K, Pajak T, Rosenthal DI, et al.: A phase III trial to compare standard versus accelerated fractionation in combination with concurrent cisplatin for head and neck carcinomas (RTOG 0129): report of compliance and toxicity. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-21, S12-13, 2007.
- [Derived] Gharzai LA, Morris E, Schipper MJ, Kidwell KM, Nguyen-Tan PF, Rosenthal DI, Gillison ML, Jordan RC, Garden AS, Koyfman SA, Caudell JJ, Blakaj DM, Dunlap NE, Krempl GA, Longo JM, Jones CU, Gensheimer MF, Galloway TJ, DeMora L, Le QT, Shah JL, Suresh K, Mierzwa M. Treatment Interruption and Outcomes in Head and Neck Cancer: A Secondary Analysis of 3 Randomized Clinical Trials. JAMA Otolaryngol Head Neck Surg. 2025 Dec 4:e254203. doi: 10.1001/jamaoto.2025.4203. Online ahead of print. PMID 41343184
- [Derived] Mell LK, Shen H, Nguyen-Tan PF, Rosenthal DI, Zakeri K, Vitzthum LK, Frank SJ, Schiff PB, Trotti AM 3rd, Bonner JA, Jones CU, Yom SS, Thorstad WL, Wong SJ, Shenouda G, Ridge JA, Zhang QE, Le QT. Nomogram to Predict the Benefit of Intensive Treatment for Locoregionally Advanced Head and Neck Cancer. Clin Cancer Res. 2019 Dec 1;25(23):7078-7088. doi: 10.1158/1078-0432.CCR-19-1832. Epub 2019 Aug 16. PMID 31420360
- [Derived] Beitler JJ, Switchenko JM, Dignam JJ, McDonald MW, Saba NF, Shin DM, Magliocca KR, Cassidy RJ, El-Deiry MW, Patel MR, Steuer CE, Xiao C, Hudgins PA, Aiken AH, Curran WJ Jr, Le QT. Smoking, age, nodal disease, T stage, p16 status, and risk of distant metastases in patients with squamous cell cancer of the oropharynx. Cancer. 2019 Mar 1;125(5):704-711. doi: 10.1002/cncr.31820. Epub 2018 Dec 11. PMID 30548235
- [Derived] Wuthrick EJ, Zhang Q, Machtay M, Rosenthal DI, Nguyen-Tan PF, Fortin A, Silverman CL, Raben A, Kim HE, Horwitz EM, Read NE, Harris J, Wu Q, Le QT, Gillison ML. Institutional clinical trial accrual volume and survival of patients with head and neck cancer. J Clin Oncol. 2015 Jan 10;33(2):156-64. doi: 10.1200/JCO.2014.56.5218. Epub 2014 Dec 8. PMID 25488965
- [Derived] Nguyen-Tan PF, Zhang Q, Ang KK, Weber RS, Rosenthal DI, Soulieres D, Kim H, Silverman C, Raben A, Galloway TJ, Fortin A, Gore E, Westra WH, Chung CH, Jordan RC, Gillison ML, List M, Le QT. Randomized phase III trial to test accelerated versus standard fractionation in combination with concurrent cisplatin for head and neck carcinomas in the Radiation Therapy Oncology Group 0129 trial: long-term report of efficacy and toxicity. J Clin Oncol. 2014 Dec 1;32(34):3858-66. doi: 10.1200/JCO.2014.55.3925. Epub 2014 Nov 3. PMID 25366680

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Started | 372 | 371
Completed | 361 | 360
Not Completed | 11 | 11
Not completed — Withdrawn consent | 2 | 3
Not completed — Ineligible | 9 | 8

BASELINE CHARACTERISTICS:
Population: Eligible patients who did not withdraw consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin | Total
Number analyzed (Participants) | 361 | 360 | 721
Age, Continuous [Median (Full Range); unit: years] | 56 [34 to 82] | 55 [26 to 82] | 56 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 72 | 124
  Male | 309 | 288 | 597

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (Percentage of Participants Alive)
Description: Overall survival time is defined as time from randomization to the date of death (failure) or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. The full distribution is the outcome of interest, and the protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year estimates are provided as a summary of the distributions. Analysis was planned to occur after 309 deaths had been reported.
Time Frame: From randomization to last follow-up. Follow-up schedule from end of treatment: 6-8 weeks, every 3 mo. for 2 yr., then every 6 mo. for 3 yr., then yearly. Maximum follow-up at time of analysis was 6.5 years. Three-year rates are reported here.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 361 | 360
percentage of patients | 64.3 [59.3 to 69.2] | 70.3 [65.6 to 75.1]
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; A sample size of 684 analyzable patients provides 80% power to detect a relative reduction of 25% in the rate of death in the accelerated-fractionation radiotherapy group as compared with the standard-fractionation radiotherapy group, assuming a 2-year rate of overall survival of 45% in the standard-fractionation radiotherapy group, with the use of a one-sided log-rank test at the 0.05 significance level; Test type: Superiority or Other; p = 0.180, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.719 to 1.128]

2. Secondary Outcome: Local-regional Failure (Percentage of Participants With Local-regional Failure)
Description: Local-regional failure time is defined as time from randomization to persistent disease in the primary tumor or regional nodes (considered an event at day 1), relapse/progression in either of those sites (considered an event at the time of relapse/progression), death (competing event), or last follow-up (censored). Progression is defined as an estimated increase in the size of the tumor of greater than 25% or appearance of new areas of malignant disease. The full distribution is the outcome of interest, and the protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year estimates are provided as a summary of the distributions. Analysis was planned to occur after 309 deaths had been reported.
Time Frame: as for outcome 1
Population: Eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 361 | 360
percentage of participants | 25.5 [21.0 to 30.0] | 28.7 [24.0 to 33.4]
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; Test type: Superiority; p = 0.76, Gray's test — One-sided significance level = 0.05; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.83 to 1.43]

3. Secondary Outcome: Local-regional Failure (Alternate Definition) [Percentage of Participants With Local-regional Failure]
Description: Local-regional failure time is defined as time from randomization to relapse/progression in the primary tumor or regional nodes (event), death due to study cancer or unknown causes (event), death due to other causes (competing event), distant metastasis (competing event), or last follow-up (censored). Progression is defined as an estimated increase in the size of the tumor of greater than 25% or appearance of new areas of malignant disease. The full distribution is the outcome of interest, and the protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year estimates are provided as a summary of the distributions. Analysis was planned to occur after 309 deaths had been reported.
Time Frame: as for outcome 1
Population: Eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 361 | 360
percentage of participants | 25.6 [21.1 to 30.1] | 28.2 [23.6 to 32.9]
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; Test type: Superiority; p = 0.80, Gray's test — One-sided significance level = 0.05; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.85 to 1.44]

4. Secondary Outcome: Disease-free Survival (Percentage of Participants Alive Without Disease)
Description: Disease-free survival time is defined as time from randomization to persistent disease in the primary tumor or regional nodes (considered an event at day 1), relapse/progression in either of those sites (considered an event at the time of relapse/progression), distant metastasis (event), second primary tumor (event), death (event), or last follow-up (censored). Progression is defined as an estimated increase in the size of the tumor of greater than 25% or appearance of new areas of malignant disease. The full distribution is the outcome of interest, and the protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year estimates are provided as a summary of the distributions. Analysis was planned to occur after 309 deaths had been reported.
Time Frame: as for outcome 1
Population: Eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 361 | 360
percentage of participants | 51.4 [46.3 to 56.6] | 53.4 [48.2 to 58.6]
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; Test type: Superiority; p = 0.42, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.81 to 1.20]

5. Secondary Outcome: Progression-free Survival (Alternate Definition of Disease-free Survival) [Percentage of Participants Alive Without Progression]
Description: Progression-free survival time is defined as time from randomization to relapse/progression in the primary site or regional nodes (event), distant metastasis (event), death (event), or last follow-up (censored). Progression is defined as an estimated increase in the size of the tumor of greater than 25% or appearance of new areas of malignant disease. The full distribution is the outcome of interest, and the protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year estimates are provided as a summary of the distributions. Analysis was planned to occur after 309 deaths had been reported.
Time Frame: as for outcome 1
Population: Eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 361 | 360
percentage of participants | 55.8 [50.6 to 60.9] | 57.0 [51.8 to 62.1]
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; Test type: Superiority; p = 0.50, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.81 to 1.23]

6. Secondary Outcome: Percentage of Participants With Toxicity Grade 3 or Higher
Description: Acute radiation therapy toxicities (within 90 days from start of radiation therapy) and systemic effects at any time were scored using Common Toxicity Criteria (CTC) version 2.0. Late RT toxicities (> 90 days from start of radiation therapy) were scored by the Radiation Therapy Oncology Group (RTOG)/European Organisation for. Research and Treatment of Cancer (EORTC) criteria. Both criteria grades toxicity severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event/toxicity data.
Time Frame: From randomization to last follow-up. Follow-up schedule from end of treatment: 6-8 weeks, every 3 mo. for 2 yr., then every 6 mo. for 3 yr., then yearly. Maximum follow-up at time of analysis was 6.5 years.
Population: Eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 361 | 360
percentage of participants
  Acute | 83.7 [79.8 to 87.5] | 80.0 [75.9 to 84.1]
  Late: number analyzed (Participants) | 351 | 343
  Late | 21.1 [16.8 to 25.3] | 25.7 [21.0 to 30.3]
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; Acute toxicity; Test type: Superiority; p = 0.21, Fisher Exact — Two-side significance level = 0.05
Statistical Analysis 2: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; Late toxicity; Test type: Superiority; p = 0.18, Fisher Exact — Two-sided significance level = 0.05

7. Secondary Outcome: Performance Status Scale for Head and Neck Cancer (PSS-HN) Normalcy of Diet Score - Area Under the Curve (AUC) at One Year
Description: The PSS-HN is a clinician-rated evaluation conducted as an unstructured interview format that assesses three functions: Normalcy of Diet (this outcome measure), Public Eating, and Understandability of Speech. Each function is scored from 0 to 100 and analyzed separately. Higher scores indicate better performance status. Treatment effect was analyzed as time-weighted average between baseline (pre-treatment) and one year calculated by use of area under the curve (AUC).
Time Frame: Baseline (pretreatment), sometime during the last two weeks of treatment, three months from start of treatment, and one year from start of treatment.
Population: Eligible patients who did not withdraw consent, with all 4 assessments: baseline, last 2 weeks of treatment, 3 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale * months
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 141 | 140
score on a scale * months | 53.36 (1.99) | 53.63 (1.97)
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; Two hundred and fifty-two patients (126/arm) provide at least 86% power to detect a difference of 7 (standard deviation 18) between arms with a two-sided significance level of 0.05; Test type: Superiority; p = 0.92, t-test, 2 sided — Two-sided significance level = 0.05

8. Secondary Outcome: PSS-HN Public Eating Score - AUC at One Year
Description: The Performance Status Scale for Head and Neck Cancer (PSS-HN) is a clinician-rated evaluation conducted as an unstructured interview format that assesses three functions: Normalcy of Diet , Public Eating (this outcome measure), and Understandability of Speech. Each function is scored from 0 to 100 and analyzed separately. Higher scores indicate better performance status. Treatment effect was analyzed as time-weighted average between baseline (pretreatment) and one year calculated by use of area under the curve (AUC).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale * months
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 126 | 131
score on a scale * months | 65.81 (2.18) | 67.10 (2.12)
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.67, t-test, 2 sided — Two-sided significance level = 0.05

9. Secondary Outcome: PSS-HN Understandability of Speech Score - AUC at One Year
Description: The Performance Status Scale for Head and Neck Cancer (PSS-HN) is a clinician-rated evaluation conducted as an unstructured interview format that assesses three functions: Normalcy of Diet , Public Eating, and Understandability of Speech (this outcome measure). Each function is scored from 0 to 100 and analyzed separately. Higher scores indicate better performance status. Treatment effect was analyzed as time-weighted average between baseline (pretreatment) and one year calculated by use of area under the curve (AUC).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale * months
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 142 | 145
score on a scale * months | 90.48 (1.18) | 91.77 (1.11)
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.43, t-test, 2 sided — Two-sided significance level = 0.05

10. Secondary Outcome: Head and Neck Radiotherapy Questionnaire (HNRQ) - AUC at One Year
Description: The HNRQ is a patient-reported questionnaire administrated through a paper format; it measures radiation-related side effects and the overall well-being of head and neck cancer patients in the past week. The overall score is the mean of the 22 questions, with a range of 1 to 7. Higher scores indicate better quality of life. Treatment effect was analyzed as time-weighted average between baseline (pre-treatment) and 1 year calculated by use of area under the curve (AUC).
Time Frame: as for outcome 7
Population: Eligible participants who did not withdraw consent, with all 4 assessments: baseline, last 2 weeks of treatment, 3 months, and one year.
Measure: Mean (Standard Error); unit: score on a scale * months
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 139 | 137
score on a scale * months | 5.27 (0.07) | 5.19 (0.07)
Statistical Analysis 1: Comparison: Standard Fractionation RT + Cisplatin vs Accelerated Fractionation RT + Cisplatin; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.39, t-test, 2 sided — Two-sided significance level = 0.05

11. Secondary Outcome: Correlation of Epidermal Growth Factor Receptor(EGFR) With Outcomes
Time Frame: From randomization to date of death or last follow-up
Population: No assays were performed and no data were collected for this outcome measure.
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Correlation of COX-2 With Outcomes
Time Frame: From randomization to date of death or last follow-up
Population: No assays were performed and no data were collected for this outcome measure.
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE).
Arm/Group | Standard Fractionation RT + Cisplatin | Accelerated Fractionation RT + Cisplatin
Serious Adverse Events (participants affected / at risk) | 293/361 | 279/360
Other Adverse Events (participants affected / at risk) | 360/361 | 356/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Fractionation RT + Cisplatin (N=361) | Accelerated Fractionation RT + Cisplatin (N=360)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 17
Hemoglobin decreased (Blood and lymphatic system disorders) | 33 | 24
Lymphatics-Other (Blood and lymphatic system disorders) | 1 | 0
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 7 | 7
Circulatory or cardiac-Other (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Endocrine-Other (Endocrine disorders) | 1 | 0
Diarrhea NOS (Gastrointestinal disorders) | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 82 | 76
Esophageal spasm (Gastrointestinal disorders) | 37 | 31
Esophagitis NOS (Gastrointestinal disorders) | 30 | 48
GI-other (Gastrointestinal disorders) | 3 | 2
Hematemesis (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0
Late RT Toxicity: Esophagus: NOS (Gastrointestinal disorders) | 28 | 37
Late RT Toxicity: Larynx: NOS (Gastrointestinal disorders) | 14 | 18
Late RT Toxicity: Mucous Membrane: NOS (Gastrointestinal disorders) | 3 | 11
Late RT Toxicity: Other: dysphagia (Gastrointestinal disorders) | 1 | 0
Late RT Toxicity: Other: tongue edema (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 72 | 52
Pancreatitis NOS (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Radiation mucositis (Gastrointestinal disorders) | 141 | 117
Salivary gland disorder NOS (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 7 | 2
Stomatitis/pharyngitis for BMT (Gastrointestinal disorders) | 1 | 0
Tracheo-oesophageal fistula NOS (Gastrointestinal disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 66 | 42
Fatigue (General disorders) | 1 | 3
Late RT Toxicity: Other: pain (General disorders) | 1 | 0
Pain due to radiation (General disorders) | 30 | 31
Pain-other (General disorders) | 9 | 7
Culture wound positive (Infections and infestations) | 0 | 2
Implant infection (Infections and infestations) | 2 | 0
Infection NOS (Infections and infestations) | 13 | 8
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 5 | 13
Infection with unknown ANC (Infections and infestations) | 0 | 2
Infection, Other (Infections and infestations) | 4 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 29 | 31
Late RT Toxicity: Subcutaneous Tissue (within XRT field): NOS (Injury, poisoning and procedural complications) | 2 | 3
Blood alkaline phosphatase NOS increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 16 | 10
Cardiac troponin T increased (Investigations) | 1 | 0
Leukopenia NOS (Investigations) | 14 | 13
Lymphopenia (Investigations) | 0 | 1
Metabolic-Other (Investigations) | 2 | 0
Neutropenia (Investigations) | 17 | 14
Platelet count decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 27 | 22
Blood magnesium decreased (Metabolism and nutrition disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 76 | 67
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 13 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | 2
Hypernatremia (Metabolism and nutrition disorders) | 3 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 3 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 3
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 28 | 17
Hyponatremia (Metabolism and nutrition disorders) | 41 | 33
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 4
Joint, muscle, or bone-Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Late RT Toxicity: Bone: NOS (Musculoskeletal and connective tissue disorders) | 14 | 18
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia NEC (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dizziness (exc vertigo) (Nervous system disorders) | 4 | 1
Headache NOS (Nervous system disorders) | 2 | 2
Hemorrhagic stroke (Nervous system disorders) | 0 | 1
Late RT Toxicity: Brain: NOS (Nervous system disorders) | 1 | 1
Late RT Toxicity: Spinal Cord: NOS (Nervous system disorders) | 0 | 1
Neurologic-Other (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 5 | 3
Vasovagal attack (Nervous system disorders) | 1 | 1
Renal failure NOS (Renal and urinary disorders) | 2 | 1
Renal/GU-Other (Renal and urinary disorders) | 7 | 3
Urinary retention (Renal and urinary disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Late RT Toxicity: Other: airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Late RT Toxicity: Other: laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Late RT Toxicity: Other: pharyngeal bleed (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Late RT Toxicity: Other: stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Late RT Toxicity: Other: upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hemorrhage-Other (Vascular disorders) | 1 | 2
Hypertension NOS (Vascular disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 6 | 7
Late RT Toxicity: Other: arteritis (Vascular disorders) | 0 | 1
Thrombosis NOS (Vascular disorders) | 2 | 1
Visceral arterial ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Fractionation RT + Cisplatin (N=361) | Accelerated Fractionation RT + Cisplatin (N=360)
Hemoglobin decreased (Blood and lymphatic system disorders) | 325 | 301
Hearing impaired (Ear and labyrinth disorders) | 63 | 35
Hearing-Other (Ear and labyrinth disorders) | 52 | 53
Constipation (Gastrointestinal disorders) | 73 | 54
Diarrhea NOS (Gastrointestinal disorders) | 37 | 27
Dry mouth (Gastrointestinal disorders) | 184 | 156
Dysphagia (Gastrointestinal disorders) | 112 | 94
Esophageal spasm (Gastrointestinal disorders) | 58 | 52
Esophagitis NOS (Gastrointestinal disorders) | 118 | 101
Late RT Toxicity: Esophagus: NOS (Gastrointestinal disorders) | 145 | 152
Late RT Toxicity: Larynx: NOS (Gastrointestinal disorders) | 161 | 132
Late RT Toxicity: Mucous Membrane: NOS (Gastrointestinal disorders) | 143 | 147
Late RT Toxicity: Salivary Gland (xerostomia, taste impairment) (Gastrointestinal disorders) | 270 | 271
Nausea (Gastrointestinal disorders) | 210 | 197
Radiation mucositis (Gastrointestinal disorders) | 282 | 267
Salivary gland disorder NOS (Gastrointestinal disorders) | 120 | 116
Stomatitis (Gastrointestinal disorders) | 29 | 19
Vomiting NOS (Gastrointestinal disorders) | 140 | 131
Edema NOS (General disorders) | 14 | 19
Fatigue (General disorders) | 212 | 198
Late RT Toxicity: Other: NOS (General disorders) | 173 | 171
Pain due to radiation (General disorders) | 144 | 135
Pain-other (General disorders) | 46 | 41
Pyrexia (General disorders) | 31 | 33
Infection NOS (Infections and infestations) | 21 | 30
Infection, Other (Infections and infestations) | 20 | 14
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 236 | 213
Late RT Toxicity: Skin(within RT field): NOS (Injury, poisoning and procedural complications) | 145 | 145
Late RT Toxicity: Subcutaneous Tissue (within XRT field): NOS (Injury, poisoning and procedural complications) | 159 | 171
Alanine aminotransferase increased (Investigations) | 32 | 34
Aspartate aminotransferase increased (Investigations) | 27 | 29
Blood alkaline phosphatase NOS increased (Investigations) | 27 | 13
Blood creatinine increased (Investigations) | 122 | 85
Leukopenia NOS (Investigations) | 302 | 254
Lymphopenia (Investigations) | 48 | 42
Metabolic-Other (Investigations) | 26 | 28
Neutropenia (Investigations) | 227 | 176
Platelet count decreased (Investigations) | 103 | 87
Weight decreased (Investigations) | 171 | 153
Anorexia (Metabolism and nutrition disorders) | 95 | 72
Blood albumin decreased (Metabolism and nutrition disorders) | 79 | 64
Blood magnesium decreased (Metabolism and nutrition disorders) | 96 | 73
Dehydration (Metabolism and nutrition disorders) | 166 | 108
Hyperglycemia NOS (Metabolism and nutrition disorders) | 67 | 57
Hyperkalemia (Metabolism and nutrition disorders) | 47 | 24
Hypocalcemia (Metabolism and nutrition disorders) | 71 | 51
Hypokalemia (Metabolism and nutrition disorders) | 84 | 67
Hyponatremia (Metabolism and nutrition disorders) | 126 | 92
Joint, muscle, or bone-Other (Musculoskeletal and connective tissue disorders) | 20 | 18
Late RT Toxicity: Bone: NOS (Musculoskeletal and connective tissue disorders) | 24 | 29
Late RT Toxicity: Joint: NOS (Musculoskeletal and connective tissue disorders) | 48 | 59
Late RT Toxicity: Spinal Cord: NOS (Nervous system disorders) | 15 | 20
Peripheral sensory neuropathy (Nervous system disorders) | 55 | 29
Taste disturbance (Nervous system disorders) | 114 | 117
Depression NEC (Psychiatric disorders) | 21 | 20
Insomnia NEC (Psychiatric disorders) | 21 | 17
Renal/GU-Other (Renal and urinary disorders) | 40 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 33
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 75 | 55
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 15
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 20 | 21
Skin-Other (Skin and subcutaneous tissue disorders) | 27 | 12

LIMITATIONS AND CAVEATS:
Local-regional failure and disease-free survival were additionally analyzed with the definition of failure used in the Meta-Analysis of Radiotherapy in Carcinomas of Head and Neck (MARCH) Collaborative Group and the Meta-Analysis of Chemotherapy in Head and Neck Cancer (MACH-NC) Collaborative Group publications. These modified outcome measures are labeled "Alternate Definition".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.